CLINICAL TRIAL: NCT02760875
Title: Foot Pressure Mapping and Ultrasound Achilles Tendon Length, in Medium Term Acute Achilles Tendon Rupture Patients Using Nonoperative Treatment.
Brief Title: Foot Pressure Mapping and Tendon Length After Nonoperative Treatment of Acute Achilles Tendon Rupture
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Rasmus Kastoft, Research Assistant, Copenhagen University Hospital, Hvidovre
Other Study IDs: 16015461-2
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles Tendon Rupture; Conservative treatment; early weight bearing; Achilles Tendon Length; Ultrasound; Foot Pressure Mapping; ATRA; Heel Raise Work

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Early Weight Bearing: Ankle immobilized with orthosis (DJO Nextep Contour 2 Walker) with 3 1.5 cm wedges in the heel, fixing the angle between 20-30 degrees. The orthosis was used for 8 weeks, gradually removing the wedges. Full weight bearing was allowed from day 1. The orthosis was worn 24 hours / day the first 2 weeks.
  From week 2 controlled motion exercises and removal of the orthosis 5 times a day.
  Interventions: Behavioral: Early weight bearing
- control: Ankle immobilized with orthosis (DJO Nextep Contour 2 Walker) with 3 1.5 cm wedges in the heel, fixing the angle between 20-30 degrees. The orthosis was used for 8 weeks, gradually removing the wedges. Full weight bearing was allowed from week 6. The orthosis was worn 24 hours / day the first 2 weeks.
  From week 2 controlled motion exercises and removal of the orthosis 5 times a day.

INTERVENTIONS:
Behavioral: Early weight bearing — The intervention implies that the selected patients, will be allowed to bear weight on the injured leg form day 1 while wearing the orthosis, in contrast to the control group, who must wait 6 weaks.
  Groups: Early Weight Bearing

SUMMARY:
Using a population of patients from another study, who was originally randomized to 2 different types of nonoperative treatment after an acute achilles tendon rupture, the length of the achilles tendon is examined using ultrasound, and foot pressure mapping is performed, 4-5 years after the injury.

DETAILED DESCRIPTION:
A total of 56 patients from an earlier study (see reference) on Achilles tendon rupture using nonoperative treatment with or without early weight bearing was invited for an additional follow up, where we examine the length of the Achilles tendon using ultrasound, as well as functional influence of the injury, using foot pressure mapping (FPM) during barefoot gait. Additionally the mobility of the ankle is measured with the Achilles Tendon Resting Angle (ATRA) as well as passive plantar- and dorsiflexion. Strength is measured using Heel Raise Work (height of lift, number of lifts and the total work), and supplemented with calf circumference.

ELIGIBILITY:
Inclusion Criteria:

* Suffered acute Achilles tendon rupture from April 2011 to March 2012, and then referred to Copenhagen University Hospital Hvidovre.
* Participated and completed the original study.
* The patient must be able to speak and understand Danish, as well as be capable to give informed consent to participating.

Exclusion Criteria:

* Terminal disease or serious illnesses with an ASA score of 3 or above.
* Any injury significantly influencing gate and function of the lower extremities other than re-rupture of the Achilles tendon.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who participated and completed the original study:
  Barfod, K.W., et al., Nonoperative dynamic treatment of acute achilles tendon rupture: the influence of early weight-bearing on clinical outcome: a blinded, randomized controlled trial. J Bone Joint Surg Am, 2014. 96(18): p. 1497-503.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Achilles Tendon Length | Test is performed once, 4-5 years after the initial injury

SECONDARY OUTCOMES:
Foot pressure mapping | Test is performed once, 4-5 years after the initial injury
  Using a pressure sensitive plate, the force excerted on the floor while walking is meassured for each part of the food (such as big toe, midfoot and heel), and data is presentred in the form of peak pressure, pressure/time integral, first contact (time) and last contact (time) for each region of the foot.
ATRA: Achilles Tendon Resting Angle | Test is performed once, 4-5 years after the initial injury.
  With the subject lying face down and the knee bent to 90 degrees, the angle between the longitudinal fibular axis and the axis of the 5. metatarsal is meassured in a relaxed state using a goniometer.
Passive plantar- and dorsiflextion | Test is performed once, 4-5 years after the initial injury
  Using a goniometer, and performed with the patient lying face down, the maximal angle that the ankle can be pushed into, while the patient is relaxing is meassured, both in regard to plantar and dorsiflexion.
circumference of the calf | Test is performed once, 4-5 years after the initial injury
  With the patient sitting on the side of the bench, the circumference of the calf is meassured 13 cm below the distal part of the kneecap.
Heel Raise Work | Test is performed once, 4-5 years after the initial injury
  The total work (joules), max height of lift (mm) and number of lifts is recorded. THe patient is placed standing on one leg on a platform tilted 10 degrees (heel below toes), and is asked to lift the heel (and thereby bodyweight) as high as possible, once every 2 seconds. When the patient can no longer maintain height or pace, the test is finished.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Penny, MD, PhD, Study Director — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barfod KW, Bencke J, Lauridsen HB, Ban I, Ebskov L, Troelsen A. Nonoperative dynamic treatment of acute achilles tendon rupture: the influence of early weight-bearing on clinical outcome: a blinded, randomized controlled trial. J Bone Joint Surg Am. 2014 Sep 17;96(18):1497-503. doi: 10.2106/JBJS.M.01273. PMID 25232073